CLINICAL TRIAL: NCT04119258
Title: Therapist Adherence to Evidence-based Cognitive-behavioral Therapy in a Patient Perspective
Brief Title: Therapist Adherence to Cognitive-behavioral Therapy
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Benjamin Bohman, Principal Investigator, Karolinska Institutet
Other Study IDs: KI-2019-04255
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Depression; Anxiety Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Psychiatric patients: Psychiatric outpatient care patients with major depressive disorder, anxiety disorders, post-traumatic stress disorder, obsessive-compulsive disorder, or illness anxiety disorder who have just completed cognitive-behavioral therapy.
  Interventions: Behavioral: Cognitive-behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy — Cognitive-behavioral therapy including both behavioral and cognitive interventions.

SUMMARY:
An observational web-based survey on therapist adherence to evidence-based cognitive-behavioral therapy (CBT) in the perspective of their patients with depression or anxiety disorders in psychiatric outpatient care in Stockholm, Sweden. Following completion of CBT, participants respond to questions including their age, gender, education, whether they have improved, whether they considered treatment helpful, and an instrument measuring therapist adherence to CBT procedures (e.g., setting agenda, follow up on home assignments) and CBT techniques (e.g., exposure, cognitive restructuring). The purpose of the study is to contribute to quality assurance of CBT in Stockholm Health Care Services.

ELIGIBILITY:
Inclusion Criteria:

* A primary diagnosis of major depressive disorder, social anxiety disorder, panic disorder, agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, post-traumatic stress disorder, or illness anxiety disorder
* 18 years of age or older
* Just completed individual cognitive-behavioral therapy in psychiatric outpatient care in Stockholm, Sweden

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psychiatric outpatient care sample
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Adherence to Cognitive-Behavioral Therapy Scale - Patient Version | Up to 20 weeks
  Patients rate the degree to which therapists adhere to evidence-based cognitive-behavioral therapy procedures and techniques on a Likert-type scale from 0 (Not at all) to 4 (To a very high degree)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Bohman, Principal Investigator — Karolinska Institutet
Locations (1):
- WeMind Psykiatri AB, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No